CLINICAL TRIAL: NCT00331877
Title: A Proactive Communication Strategy for Family Members of Patients Dying in the ICU: A Multicenter Randomized Controlled Trial
Brief Title: A Communication Strategy for Families of Patients Dying in the ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Famirea Study Group (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: famirea VIII
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2006-05-31 (Estimated); Status verified 2006-05

CONDITIONS: Family of Dying Patient in the ICU
Keywords: family; end-of-life; intensive care unit
MeSH Terms: conditions — Death

INTERVENTIONS:
Procedure: family conference with bereavement information leaflet

SUMMARY:
Decisions to limit life sustaining treatments are made for most patients dying in the ICU, usually with input from the family. The well-being of the family may be jeopardized by involvement in the decision-making process and bereavement. We evaluated the ability of a proactive communication strategy (family conference and providing family members with a bereavement information leaflet) designed to improve family well-being.

ELIGIBILITY:
Inclusion Criteria:

* family of dying patient

Exclusion Criteria:

* family having no enough knowledge of French to respond to telephone interview
* patient alive on day 90

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136
Dates: Start 2005-05; Study Completion 2006-01

PRIMARY OUTCOMES:
symptoms related to posttraumatic stress disorder

SECONDARY OUTCOMES:
symptoms of anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Elie Azoulay, Md, PhD, Study Director — Famirea Study Group

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350
- [Derived] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907